CLINICAL TRIAL: NCT05472792
Title: Comparison of Adjuvant Monotherapy With Endocrine Therapy or Accelerated Partial Breast Irradiation Following Lumpectomy for Low Risk Breast Cancer Patients Over 65 (CAMERAN)
Brief Title: Compare Adjuvant Monotherapy With Endocrine or Accelerated Partial Breast Irradiation After Lumpectomy
Acronym: CAMERAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2104-DCT
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Quality of Life
Keywords: Radiation Therapy; Endocrine Therapy; Partial Breast Irradiation; Elderly; Health Related Quality of Life; Patient Reported Outcomes
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole; exemestane; Letrozole; Fulvestrant; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Endocrine Therapy (Active Comparator): Endocrine therapy will be chosen by the treating medical oncologist with an aim of 5 years duration, as tolerated by the patient.
  Interventions: Drug: tamoxifen, anastrozole, exemestane, letrozole, fulvestrant, toremifene
- Accelerated Partial Breast Irradiation (APBI) (Experimental): APBI will consist of 5 fractions of radiation therapy delivered every other day to the lumpectomy cavity.
  Interventions: Radiation: Accelerated Partial Breast Irradiation (APBI)

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation (APBI) — Radiation treatment delivered to the lumpectomy cavity.
  Arms: Accelerated Partial Breast Irradiation (APBI)
Drug: tamoxifen, anastrozole, exemestane, letrozole, fulvestrant, toremifene — Adjuvant endocrine therapy (tamoxifen, anastrozole, exemestane, letrozole, fulvestrant, toremifene) for duration of 5 years, as tolerated by the patient.
  Arms: Endocrine Therapy

SUMMARY:
The aim of this prospective study is to investigate quality of life and oncologic outcomes in low-risk elderly breast cancer patients randomized to adjuvant therapy with accelerated partial breast irradiation (APBI) alone or endocrine therapy alone after lumpectomy. The study population will include women age 65 years and older with low-risk tumor characteristics (tumor size <2cm, grade 1-2, node-negative). APBI will consist of 5 fractions of radiation therapy delivered every other day to the lumpectomy cavity. Endocrine therapy will be chosen by the treating medical oncologist with an aim of 5 years duration, as tolerated by the patient. Quality of life outcomes will be measured at 1 year following lumpectomy and compared between groups. We hypothesize that the use of APBI may be superior in terms of quality of life when compared to endocrine therapy alone following lumpectomy while providing equivalent rates of disease control and overall survival. In this phase II study, we anticipate enrolling 90 women at N.C. Cancer Hospital in Chapel Hill, NC.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
2. Women greater than or equal to age 65 years with de novo invasive carcinoma of breast.
3. Pathological T1 (pT1) stage
4. Estrogen receptor (ER)/ Progesterone receptor (PR) positive (greater than or equal to 10% ER and PR by immunohistochemistry [IHC] staining)
5. Human epidermal growth factor receptor 2 (HER2) - according to American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) guidelines (0 or 1+ following IHC staining or proven negative by in-situ hybridization [ISH])
6. Grade 1 or 2 overall tumor grade
7. Clinical or pathological N0
8. No lymphovascular space invasion (LVSI)
9. Final surgical margins ≥ 2 mm as per APBI criteria
10. Subjects with completed breast conserving surgery (BCS) with or without sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND).
11. Suitable for APBI as deemed by the treating radiation oncologist
12. Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. Enrollment in another clinical trial is allowed if there would be no interference with interventions on this trial

Exclusion Criteria:

1. Pre- or post-operative systemic chemotherapy while on this study.
2. Current ongoing treatment with anti-hormonal agents. If previously on anti-hormonal agents and planning to stop, the subject must discontinue within 30 days of randomization.
3. Hormonal replacement therapy (eligible if discontinued within 30 days of randomization).
4. Multifocal or multicentric tumor.
5. Receipt of tissue rearrangement in the lumpectomy cavity.
6. Synchronous bilateral breast cancer.
7. Clinical or imaging evidence of distant metastases.
8. Prior breast or thoracic radiation.
9. Autoimmune conditions with associated radiation risks.
10. Subjects with poor medical risk due to uncontrolled medical conditions that would deem them ineligible for hormonal or radiation therapy.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2032-04-15 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 | 1 year
  To compare quality of life at 1 year after breast conserving surgery in those who receive adjuvant accelerated partial breast irradiation alone versus adjuvant endocrine therapy alone as measured by the EORTC QLQ-C30. Raw scores are linearly converted to a 0-100 scale with higher symptom scales reflecting increased levels of symptom burden.
Patient reported outcomes assessed by EORTC QLQ-BR45 | 1 year
  To compare quality of life at 1 year after breast conserving surgery in those who receive adjuvant accelerated partial breast irradiation alone versus adjuvant endocrine therapy alone as measured by the EORTC QLQ-BR45. Raw scores are linearly converted to a 0-100 scale with higher symptom scales reflecting increased levels of symptom burden.

SECONDARY OUTCOMES:
Disease-free survival | 2 years
  To assess the 2-year outcome of disease-free survival, including DCIS (DFS-DCIS), in subjects who have received accelerated partial breast irradiation alone versus endocrine therapy alone after breast conserving surgery
Overall survival | 2 years
  To assess the 2-year overall survival (OS) in subjects who have received accelerated partial breast irradiation alone versus endocrine therapy alone after breast conserving surgery

OTHER OUTCOMES:
Endocrine therapy adherence | 5 years
  To measure the adherence to the planned endocrine therapy in the endocrine therapy alone arm using a medication usage questionnaire
Disease-free survival | 5 years
  To assess 5-year DFS-DCIS in subjects who have received accelerated partial breast irradiation alone versus endocrine therapy alone after breast conserving surgery.
Overall survival | 5 years
  To assess 5-year OS in subjects who receive accelerated partial breast irradiation alone versus endocrine therapy alone after breast conserving surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Casey, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials